CLINICAL TRIAL: NCT03806868
Title: Dietary Intervention Increasing Omega-3 Intake- Feasibility Trial
Brief Title: Dietary Intervention Increasing Omega-3 Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB00069904; P50MD010431 (NIH)
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The Intervention group will receive a voucher for ordering foods (ONLY omega-3 rich foods) weekly (4 times).
  Interventions: Other: voucher for ordering foods (ONLY omega-3 rich foods)
- Control group (Sham Comparator): The Control group will receive a voucher for ordering foods in general (any type of foods) weekly (4 times). Participants will NOT be limited to purchasing foods rich in omega-3.
  Interventions: Other: voucher for ordering foods in general (any type of foods)

INTERVENTIONS:
Other: voucher for ordering foods (ONLY omega-3 rich foods) — A voucher will be provided weekly (4 times) for ordering only omega-3 rich foods. Groceries will be delivered to participants' home weekly.
  Arms: Intervention group
Other: voucher for ordering foods in general (any type of foods) — A voucher will be provided weekly (4 times) for ordering any type of food. Groceries will be delivered to participants' home weekly.
  Arms: Control group

SUMMARY:
This Dietary Intervention is being done to evaluate the feasibility of a food voucher program and dietary counseling to increase consumption of healthy fatty acids (omega-3) in individuals with Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
The goal of this pilot intervention is to evaluate the feasibility of a food voucher program and dietary counseling to increase dietary intake of omega-3 fatty acid in individuals with COPD.

This hypothesis is based on a number of recent observations. Studies have investigated the impact of omega-3 fatty acids, especially Eicosapentaenoic acid (EPA), Docosahexaenoic acid (DHA), alfa-linolenic acid (ALA) intake in chronic diseases and show a link with decreased systemic inflammation measured by cytokines including interleukin 1 (IL-1B), interleukin 6 (IL-6), interleukin 10 (IL-10), tumoral necrosis factor alfa (TNF-α) and eicosanoids; and improved outcomes. In a large cross-sectional study of individuals with COPD, a diet rich in the omega-3 ALA was associated with lower serum TNF-α levels while a diet rich in the omega-6's LA and arachidonic acid (AA) had higher systemic inflammatory markers IL-6 and c-reactive protein (CRP). Other recent nutritional epidemiological study showed the association of greater intakes of omega-3 fatty acids with better lung function profile, but also a slower forced expiratory volume at the 1 second (FEV1) decline in the same smoker cohort.

Preliminary cross-sectional data (n=59), from the CLEAN Air study, reported that at baseline, a higher omega 3 dietary intake was linked with reduced systemic inflammation (IL-1B) and improved respiratory outcomes (a 28% decrease in the odds of COPD symptoms in moderate-severe COPD and conversely, higher omega-6 levels associated with worse outcomes, including increased dyspnea and lower lung function. These findings support the importance of implementing an intervention program to confirm there is a beneficial association between fatty acid dietary intake and reduced COPD symptoms.

To this end, the investigators propose a pilot intervention study in 20 subjects to see if the investigators can increase omega-3 dietary intake over a 4 week period. The investigators will measure self-report dietary intake of omega 3 and 6 fatty acids, as well as measure, fasting plasma fatty acid levels, before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years,
* Physician diagnosis of COPD, Global Initiative for Obstructive Lung Disease (GOLD) Stage II-IV disease with Forced -Expiratory Volume (FEV1)/ Forced Vital Capacity (FVC) <70% and FEV1 (% predicted) <80%,
* Tobacco exposure ≥ 10 pack-years
* Former smoker with an exhaled Carbon Monoxide (eCO)<=6 ppm to confirm smoking status
* No home smoking ban.
* Subjects with low omega-3 intake (EPA+DHA levels <500mg) based on data extracted from a food frequency questionnaire (FFQ) completed before the randomization.

Exclusion Criteria:

* Chronic systemic corticosteroids,
* Other chronic lung disease including asthma,
* Living in location other than home (e.g., long term care facility)
* Homeowner or occupant planning to move or change residence within study period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Change in serum omega 3 levels | Baseline, 2 weeks and 4 weeks
  Omega 3 levels in serum (mg) will be measured at each study visit.
Change in omega 3 intake | Baseline and 4 weeks
  A food frequency questionnaire will be administered at baseline and 4 weeks after randomization to estimate omega 3 intake (mg) at each study visit

SECONDARY OUTCOMES:
Change in health status as assessed by the Clinical COPD Questionnaire (CCQ) | Baseline, 2 weeks and 4 weeks
  The CCQ is a validated score to assess health status in COPD subjects. Score ranges from 0 to 6. The higher the score indicates lower health status.
Change in the Cough and Sputum Assessment Questionnaire (CASA-Q) Score | Baseline, 2 weeks and 4 weeks
  The CASA-Q will be administered at each study visit. Total score ranges from 0 to 100, with higher scores associated with fewer symptoms/less impact due to cough or sputum.
Change in Functional status (CAT) | Baseline, 2 weeks and 4 weeks
  Functional status will be assessed with the COPD assessment test (CAT). The total score is from 0 to 40. Higher scores indicate worse COPD control
Change in FEV1 percentage predicted | Baseline, 2 weeks and 4 weeks
  Pulmonary function testing will be assessed as FEV1 percentage predicted, that is FEV1, adjusted for age, height, race and sex.

CONTACTS AND LOCATIONS:
Overall Officials: NADIA NATHALIE HANSEL, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Campus, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No